CLINICAL TRIAL: NCT05681260
Title: A Randomized Trial Using a Modified COG ABFM Regimen Backbone to Investigate Capizzi Escalating Methotrexate Versus High Dose Methotrexate in Children with Newly Diagnosed T-cell Lymphoblastic Lymphoma (T-LBL)
Brief Title: Capizzi Escalating Methotrexate Versus High Dose Methotrexate in Children with Newly Diagnosed T-cell Lymphoblastic Lymphoma (T-LBL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Beijing Children's Hospital (Other); Children's Hospital of Scow University (Unknown); West China Second University Hospital (Other); Nanjing Children's Hospital (Other); Qilu Hospital of Shandong University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Tongji Hospital (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Cancer hospital of Shandong Province (Unknown); Shenzhen Children's Hospital (Other Government); Wuhan Children's Hospital (Other); Zhejiang University School of Medicine Children's Hospital (Unknown); Shanghai Children's Hospital (Other); Ruijin Hospital (Other); Second Affiliated Hospital of Anhui Medical University (Unknown); Children's Hospital of Hebei Province (Other); Cancer Hospital of Henan Province (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Qilu Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-T-LBL-2023
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: T-cell Lymphoblastic Lymphoma
Keywords: T-cell lymphoblastic lymphoma; Pediatric; Capizzi-style Methotrexate; High dose Methotrexate; bortezomib; treatment; survival; PET scan
MeSH Terms: interventions — Prednisone; Vincristine; pegaspargase; Cyclophosphamide; Daunorubicin; Mercaptopurine; Methotrexate; Dexamethasone; Doxorubicin; Vindesine; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard risk Arm A (Experimental): Any pediatric patients with newly diagnosed T-LBL Stage II to IV who achieve at least a PR at the end of Induction (EOI). Induction I followed by consolidation, Capizzi escalating methotrexate (interim maintenance) , delayed intensification and maintenance therapy. Triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin
- Standard risk Arm B (Experimental): Any pediatric patients with newly diagnosed T-LBL Stage II to IV who achieve at least a PR at the end of Induction (EOI). Induction I followed by consolidation, high dose methotrexate (interim maintenance) , delayed intensification and maintenance therapy. Triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin
- High Risk T-LBL (Experimental): Any pediatric patients with newly diagnosed T-LBL Stage II to IV who fail to achieve at least a PR at the end of Induction (EOI). Induction I followed by 6 intensive polychemotherapy blocks (HR1'-HR2'-HR3'-HR1'-HR2'-HR3'), deIayed intensification, and maintenance therapy. Triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin, Vindesine, Etoposide, Ifosfamide

INTERVENTIONS:
Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin — Standard risk Arm A: Induction I followed by Consolidation, extracompartmental Capizzi MTX, delayed intensification and 96 weeks' maintenance therapy. Twenty-one or twenty-six triple intrathecal injections for CNS negative or positive patients, respectively.
  Arms: Standard risk Arm A
Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin — Standard risk Arm B: Induction I followed by Consolidation, extracompartmental high dose MTX, delayed intensification and 96 weeks' maintenance therapy. Twenty-one or twenty-six triple intrathecal injections for CNS negative or positive patients, respectively.
  Arms: Standard risk Arm B
Drug: Prednisone,Vincristine, Pegylated-asparaginase, Bortezomib,Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine, methotrexate, Dexamethasone, Doxorubicin, Vindesine, Etoposide, Ifosfamide — High Risk T-LBL: Induction I followed by 2 cycles of BFM HR Blocks, delayed intensification and 96 weeks' maintenance therapy. Twenty-four or twenty-eight triple intrathecal injections for CNS negative or positive patients, respectively.
  Arms: High Risk T-LBL

SUMMARY:
T-cell lymphoblastic lymphoma (T-LBL) is the second most common subtype of non-Hodgkin lymphoma (NHL) in children and adolescents. With current treatment, event-free survival (EFS) rates vary between 75%~85%. Two different MTX intensification strategies are used commonly: HD-MTX with leucovorin rescue, and Capizzi-style MTX without leucovorin rescue plus PEG-ASP (C-MTX). Although superior outcome of patients with T-ALL receiving C-MTX compared with HD-MTX on the AALL0434 trial, the 2 approaches had not been compared directly in patients with T-LBL. There remains controversy on PET/CT interpretation in children with NHL. Large prospective studies in pediatric patients with T-LBL regarding PET/CT value for this is scarce. Around 1% pediatric patients with T-LBL will not achieve remission at the end of Induction (induction failure). The optimal treatment for this small subgroup is largely unclear. The BFM HR Blocks usually are applied to these patients even though the efficacy is unknown. Novel targeted therapies are needed for use. Dasatinib is identified as a targeted therapy for T-cell ALL in preclinical drug screening.

DETAILED DESCRIPTION:
1. T-cell lymphoblastic lymphoma (T-LBL) which involves 90% of LBL cases is the second most common subtype of non-Hodgkin lymphoma (NHL) in children and adolescents. With current treatment, event-free survival (EFS) rates vary between 75%~85%. Poor probabilities of survival (10~15%) for patients after relapse leave no room for treatment de-escalation in frontline protocols. Limitations in numbers of newly diagnosed patients impeded evaluation potential prognostic markers and validation or conducting clinical studies.
2. In the GER-GPOH-NHL-BFM-95 study, the prophylactic cranial radiation was omitted, and the intensity of induction therapy was decreased slightly. There were no significant increases in CNS relapses, suggesting cranial radiation may be reserved for patients with CNS disease at diagnosis. The 5-year EFS was worse in NHL-BFM-95 (82%) than in NHL-BFM-90 (90%). It was proposed that the major difference in EFS between NHL-BFM-90 and NHL-BFM-95 resulted from the increased number of subsequent neoplasms observed in NHL-BFM-95.
3. Two different MTX intensification strategies are used commonly: HD-MTX with leucovorin rescue, and Capizzi-style MTX without leucovorin rescue plus PEG-ASP (C-MTX). Although superior outcome of patients with T-ALL receiving C-MTX compared with HD-MTX on the AALL0434 trial, the 2 approaches had not been compared directly in patients with T-LBL.
4. POG 9404: the small cohort (n = 66) of lymphoma patients who did not receive HD-MTX, the 5-year EFS was 88%. Of note, all of these patients received prophylactic cranial radiation therapy, which has been demonstrated not to be required in T-cell lymphoblastic lymphoma (T-LBL) patients.
5. COG-A5971 evaluated 2 strategies for CNS prophylaxis without CNS irradiation [5]. Patients were randomly assigned to receive HD-MTX in interim maintenance (BFM-95) or intrathecal chemotherapy throughout maintenance (CCG-BFM). The overall incidence of CNS relapse was 1.2%, and there was no difference between the treatment arms for CNS relapse, DFS, or OS. Minimal disseminated disease (MDD) >1% by FLOW at diagnosis was shown to be associated with a worse outcome in this trial (a BFM backbone containing HD-MTX). Measurement of bone marrow MDD at diagnosis with sequential response monitoring through peripheral blood during remission induction to aid treatment stratification was also suggested in an early COG study. The prognostic significance of MDD at End-of-Induction (EOI) or End-of-Consolidation (EOC) for T-LBL patients with positive MDD at diagnosis is still unclear.
6. COG AALL0434: the COG ABFM regimen with C-MTX provided excellent DFS without cranial radiation for patients with standard risk T-LBL (85%, Arm A, n=82, completed 64) and high risk T-LBL (85%, Arm A, n=61, completed 51) although patients with CNS 3 were not included. It appears that C-MTX may have negated the prognostic impact of MDD.
7. Nelarabine is unavailable in mainland China at this time, which did not show benefit in COG AALL0434 study.
8. AALL07P1: 10 patients with T-LBL in first relapse treated with a 4-drug induction regimen adding bortezomib: 7 had a response (1 had a complete response, 2 had unconfirmed complete responses, and 4 had partial responses)
9. COG AALL1231 for T-LBL: the 4-year EFS and OS were better in bortezomib group than the control group (86.4% and 89.5% vs. 76.5% and 78.3%, p=0.041 and 0.009, respectively.). Incorporating bortezomib into standard therapy for de novo T-LBL appears beneficial.
10. A biopsy for pathological examination of a mediastinal residual mass is a clinical dilemma. Currently, conventional imaging is still considered as the "standard" modality for evaluating pediatric patients with NHL at diagnosis and subsequent response. There remains controversy on PET/CT interpretation in children with NHL. Large prospective studies in pediatric patients with T-LBL regarding PET/CT value for this is scarce.
11. Although an overlap in morphology and immune-phenotyping exists in T-LBL and T-cell acute lymphoblastic leukemia (T-ALL), different disease distribution suggests possible different genetic profiles and pathogenesis. Except for stage, none of other parameters is used in the current stratification system outside of clinical trials for T-LBL (several candidates, but none have been validated sufficiently). Little is known about biomarkers with prognostic relevance for T-LBL. To improve risk stratification strategy and better understand biologic rationale for incorporating novel therapies (chemicals, target agents and immunotherapy) into a conventional chemotherapy backbone, translational research to identify molecular markers with prognostic relevance in T-LBL is highly recommended.
12. With the current treatment, around 1% pediatric patients with T-LBL will not achieve remission at the end of Induction (induction failure). The optimal treatment for this small subgroup is largely unclear. The BFM HR Blocks usually are applied to these patients even though the efficacy is unknown. Novel targeted therapies are needed for use. Dasatinib is identified as a targeted therapy for T-cell ALL in preclinical drug screening.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T-lineage lymphoblastic lymphoma (T-LBL) Stage II-IV

Exclusion Criteria:

* Patients with Down syndrome or primary immune comprised disease.
* Ph+ T-LBL
* Patients must not have received any prior cytotoxic chemotherapy
* Any steroids pretreatment for > 5 days in the 7 days or for >14 days in the 28 days before the initiation of Induction chemotherapy. The dose of prednisone or methylprednisone pretreatment does not affect eligibility. Any steroids exposure that occurred > 28 days before the initiation of Induction chemotherapy is allowed. Inhalation and topical steroids are not considered pretreatment. A single dose of vincristine is allowed.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival for standard risk patients | 4 years
  To determine the EFS in patients with newly diagnosed standard T-LBL, through randomization, the modified COG ABFM regimen with CMTX to the regimen with HD MTX
Event free survival according to bone marrow MDD | 4 years
  After using the modified COG ABFM regimen, to validate whether bone marrow MDD by Flow at diagnosis is still a prognostic factor for pediatric patients newly diagnosed with T-LBL
Event free survival for high risk patients | 4 years
  To determine the EFS in patients with induction failure who become complete or partial response after using 3 HR BFM Blocks and continue chemotherapy on 3 HR BFM Blocks followed by delayed intensification and maintenance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (2):
- China (2):
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Chengdu

REFERENCES:
- [Background] Burkhardt B, Reiter A, Landmann E, Lang P, Lassay L, Dickerhoff R, Lakomek M, Henze G, von Stackelberg A. Poor outcome for children and adolescents with progressive disease or relapse of lymphoblastic lymphoma: a report from the berlin-frankfurt-muenster group. J Clin Oncol. 2009 Jul 10;27(20):3363-9. doi: 10.1200/JCO.2008.19.3367. Epub 2009 May 11. PMID 19433688
- [Background] Burkhardt B, Woessmann W, Zimmermann M, Kontny U, Vormoor J, Doerffel W, Mann G, Henze G, Niggli F, Ludwig WD, Janssen D, Riehm H, Schrappe M, Reiter A. Impact of cranial radiotherapy on central nervous system prophylaxis in children and adolescents with central nervous system-negative stage III or IV lymphoblastic lymphoma. J Clin Oncol. 2006 Jan 20;24(3):491-9. doi: 10.1200/JCO.2005.02.2707. PMID 16421426
- [Background] Winter SS, Dunsmore KP, Devidas M, Wood BL, Esiashvili N, Chen Z, Eisenberg N, Briegel N, Hayashi RJ, Gastier-Foster JM, Carroll AJ, Heerema NA, Asselin BL, Gaynon PS, Borowitz MJ, Loh ML, Rabin KR, Raetz EA, Zweidler-Mckay PA, Winick NJ, Carroll WL, Hunger SP. Improved Survival for Children and Young Adults With T-Lineage Acute Lymphoblastic Leukemia: Results From the Children's Oncology Group AALL0434 Methotrexate Randomization. J Clin Oncol. 2018 Oct 10;36(29):2926-2934. doi: 10.1200/JCO.2018.77.7250. Epub 2018 Aug 23. PMID 30138085
- [Background] Asselin BL, Devidas M, Wang C, Pullen J, Borowitz MJ, Hutchison R, Lipshultz SE, Camitta BM. Effectiveness of high-dose methotrexate in T-cell lymphoblastic leukemia and advanced-stage lymphoblastic lymphoma: a randomized study by the Children's Oncology Group (POG 9404). Blood. 2011 Jul 28;118(4):874-83. doi: 10.1182/blood-2010-06-292615. Epub 2011 Apr 7. PMID 21474675
- [Background] Termuhlen AM, Smith LM, Perkins SL, Lones M, Finlay JL, Weinstein H, Gross TG, Abromowitch M. Disseminated lymphoblastic lymphoma in children and adolescents: results of the COG A5971 trial: a report from the Children's Oncology Group. Br J Haematol. 2013 Sep;162(6):792-801. doi: 10.1111/bjh.12460. Epub 2013 Jul 24. PMID 23889312
- [Background] Coustan-Smith E, Sandlund JT, Perkins SL, Chen H, Chang M, Abromowitch M, Campana D. Minimal disseminated disease in childhood T-cell lymphoblastic lymphoma: a report from the children's oncology group. J Clin Oncol. 2009 Jul 20;27(21):3533-9. doi: 10.1200/JCO.2008.21.1318. Epub 2009 Jun 22. PMID 19546402
- [Background] Hayashi RJ, Winter SS, Dunsmore KP, Devidas M, Chen Z, Wood BL, Hermiston ML, Teachey DT, Perkins SL, Miles RR, Raetz EA, Loh ML, Winick NJ, Carroll WL, Hunger SP, Lim MS, Gross TG, Bollard CM. Successful Outcomes of Newly Diagnosed T Lymphoblastic Lymphoma: Results From Children's Oncology Group AALL0434. J Clin Oncol. 2020 Sep 10;38(26):3062-3070. doi: 10.1200/JCO.20.00531. Epub 2020 Jun 17. PMID 32552472
- [Background] Horton TM, Whitlock JA, Lu X, O'Brien MM, Borowitz MJ, Devidas M, Raetz EA, Brown PA, Carroll WL, Hunger SP. Bortezomib reinduction chemotherapy in high-risk ALL in first relapse: a report from the Children's Oncology Group. Br J Haematol. 2019 Jul;186(2):274-285. doi: 10.1111/bjh.15919. Epub 2019 Apr 7. PMID 30957229
- [Background] Teachey DT, Devidas M, Wood BL, Chen Z, Hayashi RJ, Hermiston ML, Annett RD, Archer JH, Asselin BL, August KJ, Cho SY, Dunsmore KP, Fisher BT, Freedman JL, Galardy PJ, Harker-Murray P, Horton TM, Jaju AI, Lam A, Messinger YH, Miles RR, Okada M, Patel SI, Schafer ES, Schechter T, Singh N, Steele AC, Sulis ML, Vargas SL, Winter SS, Wood C, Zweidler-McKay P, Bollard CM, Loh ML, Hunger SP, Raetz EA. Children's Oncology Group Trial AALL1231: A Phase III Clinical Trial Testing Bortezomib in Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia and Lymphoma. J Clin Oncol. 2022 Jul 1;40(19):2106-2118. doi: 10.1200/JCO.21.02678. Epub 2022 Mar 10. PMID 35271306
- [Background] Rosolen A, Perkins SL, Pinkerton CR, Guillerman RP, Sandlund JT, Patte C, Reiter A, Cairo MS. Revised International Pediatric Non-Hodgkin Lymphoma Staging System. J Clin Oncol. 2015 Jun 20;33(18):2112-8. doi: 10.1200/JCO.2014.59.7203. Epub 2015 May 4. PMID 25940716
- [Background] Sandlund JT, Guillerman RP, Perkins SL, Pinkerton CR, Rosolen A, Patte C, Reiter A, Cairo MS. International Pediatric Non-Hodgkin Lymphoma Response Criteria. J Clin Oncol. 2015 Jun 20;33(18):2106-11. doi: 10.1200/JCO.2014.59.0745. Epub 2015 May 4. PMID 25940725
- [Background] Bhojwani D, McCarville MB, Choi JK, Sawyer J, Metzger ML, Inaba H, Davidoff AM, Gold R, Shulkin BL, Sandlund JT. The role of FDG-PET/CT in the evaluation of residual disease in paediatric non-Hodgkin lymphoma. Br J Haematol. 2015 Mar;168(6):845-53. doi: 10.1111/bjh.13219. Epub 2014 Nov 10. PMID 25382494
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Teachey DT, O'Connor D. How I treat newly diagnosed T-cell acute lymphoblastic leukemia and T-cell lymphoblastic lymphoma in children. Blood. 2020 Jan 16;135(3):159-166. doi: 10.1182/blood.2019001557. PMID 31738819
- [Background] Khanam T, Sandmann S, Seggewiss J, Ruether C, Zimmermann M, Norvil AB, Bartenhagen C, Randau G, Mueller S, Herbrueggen H, Hoffmann P, Herms S, Wei L, Woeste M, Wuensch C, Gowher H, Oschlies I, Klapper W, Woessmann W, Dugas M, Burkhardt B. Integrative genomic analysis of pediatric T-cell lymphoblastic lymphoma reveals candidates of clinical significance. Blood. 2021 Apr 29;137(17):2347-2359. doi: 10.1182/blood.2020005381. PMID 33152759
- [Background] Laukkanen S, Gronroos T, Polonen P, Kuusanmaki H, Mehtonen J, Cloos J, Ossenkoppele G, Gjertsen B, Oystein B, Heckman C, Heinaniemi M, Kontro M, Lohi O. In silico and preclinical drug screening identifies dasatinib as a targeted therapy for T-ALL. Blood Cancer J. 2017 Sep 8;7(9):e604. doi: 10.1038/bcj.2017.87. No abstract available. PMID 28885610
- [Background] Steinherz PG. CNS leukemia: problem of diagnosis, treatment, and outcome. J Clin Oncol. 1995 Feb;13(2):310-3. doi: 10.1200/JCO.1995.13.2.310. No abstract available. PMID 7844591
- [Background] Salzburg J, Burkhardt B, Zimmermann M, Wachowski O, Woessmann W, Oschlies I, Klapper W, Wacker HH, Ludwig WD, Niggli F, Mann G, Gadner H, Riehm H, Schrappe M, Reiter A. Prevalence, clinical pattern, and outcome of CNS involvement in childhood and adolescent non-Hodgkin's lymphoma differ by non-Hodgkin's lymphoma subtype: a Berlin-Frankfurt-Munster Group Report. J Clin Oncol. 2007 Sep 1;25(25):3915-22. doi: 10.1200/JCO.2007.11.0700. PMID 17761975